CLINICAL TRIAL: NCT02267148
Title: Utilizing Non-Invasive Fibroscan® Technology to Identify Genetic Markers for Fatty Liver Progression
Status: Completed | Type: Observational
Sponsor: UNC Nutrition Research Institute (Other)
Responsible Party: Principal Investigator, Karen D. Corbin, PhD, RD, Research Assistant Professor, UNC Nutrition Research Institute
Other Study IDs: 13-1392
Record Dates: First submitted 2014-09-22; First posted 2014-10-17 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Non-alcoholic fatty liver disease; Fatty liver; Steatosis; Fibrosis; Liver Stiffness; Cirrhosis; Genetics; Single Nucleotide Polymorphism
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood will be collected and used for DNA extraction. Plasma and serum will also be collected and banked.
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a common disorder, affecting ~30% of people in the general population and up to 96% of obese individuals. Variations in several genes have been found to be associated with fatty liver, but these associations only explain a small percentage of the risk, and further studies are needed. In many cases NAFLD does not cause serious side effects, but in some individuals it progresses to scarring or hardening of the liver, liver failure, and cancer.

The purpose of this research study is to determine if individuals who carry certain genetic variations in a gene related to bile and choline metabolism have an increased risk of fatty liver progressing to fibrosis, or scarring of the liver. This study will also use a new, non-invasive method called the FibroScan® to measure liver fat and liver stiffness. The FibroScan® device is FDA approved for use to measure liver stiffness, but not for the liver fat measurement. However, the FibroScan® instrument is considered a non-significant risk device. Since its induction in Europe and worldwide in 2003, there have been no adverse effects reported with this device.

DETAILED DESCRIPTION:
Purpose: ABCB4 is a gene that intersects choline and bile metabolism, two processes that are highly relevant for liver disease. The investigators have identified a pattern of genetic variation that is associated with fatty liver burden and potentially, risk for liver disease. One of the most prominent genes in this pattern is ABCB4. This data needs to be replicated in the general population. This study will test the hypothesis that aberrant function of ABCB4 due to genetic variations will increase the risk of fatty liver progression to fibrosis. It will also implement innovative, non-invasive technology to measure liver fat and fibrosis utilizing the FibroScan® instrument. As additional proof of principle that the measurements we are making correlate with genetics, the investigators will also measure two genetic variants that have been shown in many studies to correlate with liver fat and fibrosis by their research team and others: PNPLA3 rs738409 and rs2281135. Finally, the investigators will calculate a NAFLD-Fibrosis score as an additional correlate to liver disease status.

Participants: To test this hypothesis, 50 ethnically diverse, overweight or obese male and female adults will be recruited from the general population.

Procedures: Genotyping to correlate variation in the ABCB4 and PNPLA3 genes with level of fatty liver and progression to fibrosis with the FibroScan®. Calculation of NAFLD-Fibrosis score.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Ages 18-70 years
* Body mass index 25-45

Exclusion Criteria:

* Alcohol consumption > 20 grams/day
* Liver disease from a cause other than NAFLD (such as hepatitis B/C, alcoholic liver disease, or autoimmune hepatitis)
* Pharmacological therapy for liver disease
* History of liver transplant
* Presence of implantable medical devices
* Ascites
* Pregnancy
* Smoking or use of recreational drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of the greater Charlotte, NC metropolitan area
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Liver stiffness measurement via transient elastography | Study Day 1
  Measured by FibroScan® instrument
Liver fat measurement via Controlled Attenuation Parameter | Study Day 1
  Measured using FibroScan® instrument

SECONDARY OUTCOMES:
NAFLD-Fibrosis score | Study Day 1
  This is a calculated score which is a good predictor of liver disease

CONTACTS AND LOCATIONS:
Overall Officials: Karen Corbin, PhD, RD, Principal Investigator — UNC Nutrition Research Institute
Locations (1):
- UNC Nutrition Research Institute, Kannapolis, North Carolina, United States